CLINICAL TRIAL: NCT04485000
Title: Online 1-Day CBT-Based Workshops for Postpartum Depression
Brief Title: Online 1-Day CBT-Based Workshops for PPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Ryan Van Lieshout, MD, PhD, MD, PhD, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONLINE1DAYCBT
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Participants and the research coordinator cannot be blinded to group condition, but staff making reminders and data analysts will not be aware of group status. Therapists delivering groups will be randomly assigned to workshops and not notified of group status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment (Experimental): The experimental (immediate workshop) group will receive the online workshop at baseline (T1) in addition to receiving standard postnatal care.
  Interventions: Behavioral: Online 1-Day Cognitive Behavioural Therapy (CBT)-Based Workshop
- Waitlist Cpntrol (Other): The waitlist control group will receive standard postnatal care for 12 weeks and will participate in the online 1-day CBT-based workshop at T2 (12 weeks post baseline).
  Interventions: Behavioral: Online 1-Day Cognitive Behavioural Therapy (CBT)-Based Workshop

INTERVENTIONS:
Behavioral: Online 1-Day Cognitive Behavioural Therapy (CBT)-Based Workshop — The workshop is a day-long intervention delivered in 4 modules based on Cognitive Behavioural Therapy (CBT). The workshop covers PPD etiology, modifiable cognitive risk factors, cognitive skills, behavioural skills, problem solving, goal setting and action planning. Each participant is given a professionally designed manual to facilitate learning. Weekly reminder emails are sent for 6 weeks after the workshop completion to encourage practice. A list of PPD resources and a copy of the Canadian Treatment Guidelines for Postpartum Depression are provided.

SUMMARY:
Postpartum depression (PPD) already affects up to 1 in 5 women and left untreated costs $150,000 per case over the lifespan. Under normal conditions, just 10% of women with PPD get evidence-based treatment, a situation that has worsened substantially during COVID-19. The purpose of this study is to a assess if self-referred, online adaptation of a 1-Day Cognitive Behavioural Therapy (CBT)-Based Workshop for PPD delivered up to 30 women at a time can lead to reductions in PPD, if the workshops are cost-effective, and to assess workshop impact on common complications of PPD (anxiety, partner relationship discord, problems with mother-infant attachment). 388 women will be randomized to receive either immediate treatment or treatment 12 weeks later (waitlist control). Study measures will be collected at baseline (immediately before treatment workshop) and 12 weeks later (immediately before wait list control workshop).

DETAILED DESCRIPTION:
The COVID-19 pandemic has further exposed the vulnerabilities in social and economic systems that lead to inequalities for mothers with mental health problems and their children, worsening unintended systematic biases that exist within the healthcare system. These women have been among the most affected by the pandemic, experiencing substantial worry, isolation, loneliness, lack of control, and insomnia (1), all of which have increased PPD rates. They also have more responsibilities than ever before, providing care to their infants, toddlers, and older children, while managing their households and supporting their partners. They are also profoundly worried about job losses, reduced income, and food insecurity , all of which have disrupted family routines, increased partner conflict, and rates of intimate partner violence (2).

Postpartum depression (PPD) typically affects up to 1 in 5 women (3-5), increasing the risk of later depressive episodes (6), parenting problems (7), poor mother-infant attachment (8), and emotional, behavioural, and school problems in offspring (9,10). A single case of PPD has been estimated to cost as much as $150,000 over the lifespan (11), or $57 billion for each annual cohort of Canadian births. Even under ideal conditions, the healthcare system is poorly equipped to provide care for problems requiring urgent psychotherapy like PPD (e.g., just 1 in 10 women with PPD receive evidence-based care) (12). Barriers to care include women's preference for psychotherapy over medication, a lack of time, and a reluctance to travel to regular appointments (13,14). The healthcare system is now even less able to help these women as public health units that previously supported the mental health of mothers have shifted their priorities to direct COVID response. Moreover, social distancing recommendations aimed at reducing COVID-19 risk have inadvertently increased psychological distress and decreased access to resources that protect against PPD including social and practical support from family, friends, and professionals. The need for safe and accessible PPD treatment is further highlighted by the uptake of recent recommendations (written by the NPI) on managing PPD during COVID-19 which have been read 40,000 times since their posting (12).

Only interventions that are considered safe and that can be rapidly upscaled can have an impact on PPD at the population level during COVID-19 (15). Ideal large-scale interventions for PPD during COVID-19 are not only safe (i.e., delivered online), but are brief, utilize the treatments most preferred by women (i.e., non-pharmacological), easily accessible (i.e., self-referred), provide skills that can be used over the long-term, and delivered in large groups to increase social support. At present time, no interventions exist that meet all of these criteria.

The purpose of this study is to assess if Online 1-Day CBT-Based Workshops for PPD added to care as usual during the COVID-19 pandemic improve PPD more than usual care alone, if the workshops are cost-effective, and if these workshops reduce the impact of the common comorbidities and complications of PPD (anxiety, partner relationship discord, and poorer mother-infant attachment).

388 women who are 18 years or older, have a baby under 1 year old and have an Edinburgh Postnatal Depression Scale (EPDS) score of 10 or more will be randomized to receive either immediate treatment or treatment 12 weeks later (waitlist control) and changes in depression, anxiety, relationship quality, and mother-infant attachment will be compared.

PPD is a major public health issue that has only increased in scope and impact during COVID-19, and no safe, accessible, scalable solutions exist to tackle the scope of this problem. Only health system interventions like ours that utilize existing infrastructure from a previous RCT of face-to-face workshop delivery can be launched expediently on a large scale to significantly improve the health of Canadian women with PPD and their families during this pandemic.

Promising data from a face-to-face trial, and very encouraging recruitment and feasibility findings from the online adaptation of these workshops suggest that self-referred Online 1-Day CBT-Based Workshops can be delivered immediately and rapidly scaled to reduce the impact of COVID-19 on women with PPD and their families. Since the pandemic will have a lasting impact on the delivery of mental healthcare, these online workshops could represent a significant component of the next successfully implemented, research-enabled Canadian public health strategy, and will be applicable globally.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* infant under 12 months old
* EPDS score 10 or more
* Fluent in written/spoken English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) | Differences between experimental and control groups from T1 (baseline) to T2 (12 weeks) will be compared.
  The gold standard measure of PPD in clinical practice/research. Produces a score of 0-30, with higher scores indicating more severe depressive symptoms. A change of 4 points is recognized as a clinically meaningful/significant improvement.

SECONDARY OUTCOMES:
Cost-effectiveness: Costs of service | Resources consumed over the 12-week trial period from the perspective of public healthcare payer will be measured.
  Healthcare resource utilization data will be collected using a questionnaire based on the Canadian Community Health Survey and the Service Use and Resources Form adapted for the postpartum period and used in previous PPD research. Costs will be calculated using provincial or other standard billing rates.
Cost-effectiveness: Quality-Adjusted Life Year (QALY) | QALYs will be measured over the 12-week trial period.
  The EQ-5D-5L, a utility-based health-related quality of life instrument will be used. Its validity in measuring the impact of depression is established. Its Canadian scoring algorithm will be used. For each participant, a QALY will be calculated by multiplying the health utility for the matching time period (i.e., the area under the curve approach).

OTHER OUTCOMES:
Generalized Anxiety Disorder-7 (GAD-7) | 12 weeks
  A 7-item self-report scale of symptoms of generalized anxiety disorder, the most common PPD comorbidity. This scale produces a total score of 21, with higher scores indicating more severe anxiety.
Postpartum Bonding Questionnaire | 12 weeks
  25-item maternal-report scale of mother-infant attachment. Maximum possible score is 125, with higher scores indicating more impaired mother-infant bonding.
Social Provisions Scale | 12 weeks
  The SPS is a 24-item self-report measures of the degree to which an individual's social relationships provide support.
Infant Behavior Questionnaire - Revised (Very Short Form) | 12 weeks
  A 37-item measure of infant behavior and temperament. The mean of the items to which a response of 1-7 was provided is taken for each subscale assessed. Responses of N/A are not included in the mean calculation.
Beck Depression Inventory-II (BDI-II) | 12 weeks
  Differences between experimental and control groups from T1 (baseline) to T2 (12 weeks) will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Van Lieshout, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Lieshout RJ, Layton H, Savoy CD, Brown JSL, Ferro MA, Streiner DL, Bieling PJ, Feller A, Hanna S. Effect of Online 1-Day Cognitive Behavioral Therapy-Based Workshops Plus Usual Care vs Usual Care Alone for Postpartum Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2021 Nov 1;78(11):1200-1207. doi: 10.1001/jamapsychiatry.2021.2488. PMID 34495285
- [Derived] Layton H, Owais S, Savoy CD, Van Lieshout RJ. Depression, Anxiety, and Mother-Infant Bonding in Women Seeking Treatment for Postpartum Depression Before and During the COVID-19 Pandemic. J Clin Psychiatry. 2021 Jul 6;82(4):21m13874. doi: 10.4088/JCP.21m13874. PMID 34232578